CLINICAL TRIAL: NCT03957733
Title: Phase II/III Randomized Multicentre Study Comparing Neoadjuvant Chemoradiotherapy Followed by Consolidation Chemotherapy to Neoadjuvant Chemoradiotherapy Alone in Non-metastatic Rectal Cancer Patients.
Brief Title: Phase II/III Study to Assess the Efficacy of Neoadjuvant Consolidation Chemotherapy in Rectal Cancer Patients.
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Abdullah Medical City (Other Government)
Collaborators: King Faisal Specialist Hospital & Research Center (Other); King Saud Medical City (Other Government); Al Hada Military Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-329
Record Dates: First submitted 2019-05-01; First posted 2019-05-21 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Drug Therapy; Folfox protocol; XELOX

STUDY DESIGN:
Intervention Model Description: Phase II/III randomized controlled parallel group study. Patients are randomized between Chemoradiotherapy followed by surgery or chemoradiotherapy followed by folfox/xelox chemotherapy then surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): Long course CRT is followed by 4 cycles of combination chemotherapy of modified FOLFOX6 or 3 cycles of XELOX (capecitabine and oxaliplatin) and surgery. Consolidation chemotherapy will start 2-4 weeks after the end of CRT. Surgery will be performed 2-4 weeks after the last chemotherapy cycle. After surgery, patients with pT0-2 N0 will not receive adjuvant chemotherapy. Patients with higher pathological stage will receive adjuvant chemotherapy (4 cycles of modified FOLFOX6 or 3 cycles of XELOX).
  Interventions: Drug: Chemotherapy
- Standard arm (No Intervention): Long course CRT will be followed by surgery 10-12 weeks after the end of CRT. After surgery, patients with pT0-2 N0 will not receive adjuvant chemotherapy. Patients with higher pathological stage will receive adjuvant chemotherapy (8 cycles of modified FOLFOX6 or 6 cycles of XELOX).

INTERVENTIONS:
Drug: Chemotherapy — Long course CRT is followed by 4 cycles of combination chemotherapy of modified FOLFOX6 or 3 cycles of XELOX (capecitabine and oxaliplatin) and then surgery
  Other Names: Folfox; Xelox
  Arms: Experimental arm

SUMMARY:
This is a Phase II/III randomized study involving non-metastatic rectal cancer patients who are candidates for neoadjuvant chemoradiotherapy. Eligible patients will be randomized between two treatment arms:

Experimental arm: Long course CRT is followed by 4 cycles of combination chemotherapy of modified FOLFOX6 or 3 cycles of XELOX and then surgery. After surgery, patients with pT0-2 N0 will not receive adjuvant chemotherapy. Patients with higher pathological stage will receive adjuvant chemotherapy (4 cycles of modified FOLFOX6 or 3 cycles of XELOX).

Standard arm: Long course CRT will be followed by surgery 10-12 weeks after the end of CRT. After surgery, patients with pT0-2 N0 will not receive adjuvant chemotherapy. Patients with higher pathological stage will receive adjuvant chemotherapy (8 cycles of modified FOLFOX6 or 6 cycles of XELOX).

The study aims to assess the efficacy of consolidation chemotherapy given in the interval between the end of CRT and surgery to allow for early initiation of systemic therapy aiming to decrease distant relapse rate and enhancing pathological response.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at diagnosis
* Histopathological diagnosis of rectal adenocarcinoma
* ECOG Performance Status (PS): 0- 2
* Clinical Stage: T2 N1-2, T3N0-2, T4 N0-2 based on pelvic MRI. Lymph node will be considered radiologically positive if: - size (short axis≥ 1cm) and/or - Morphological changes: irregular outlines/ abnormal signal intensity, positive enhancement.
* The standard treatment recommendation of included patients in the absence of a clinical trial would be combined modality neoadjuvant CRT followed by curative intent surgical resection.
* Primary surgeon is planning to perform Total Mesorectal Excision (TME).
* The following laboratory values must be obtained ≤ 28 days prior to registration:

  * Absolute neutrophil count (ANC) ≥ 1500/mm3
  * Platelet count ≥ 100,000/mm3
  * Hemoglobin > 8.0 g/dl (transfusion permitted)
  * Total bilirubin ≤ 1.5 x upper limit of normal (ULN)
  * SGOT (AST) ≤ 3 x ULN
  * SGPT (ALT) ≤ 3 x ULN
  * Creatinine ≤1.5 x ULN or Creatinine clearance > 50ml/minute by Cockcroft-Gault formula.
* Negative pregnancy test ≤ 7 days prior to registration for women of childbearing potential only.
* Patient of child-bearing potential is willing to employ an adequate contraception method
* Provide informed written consent
* Willing to return to the enrolling medical site for all study assessments

Exclusion Criteria:

* Extensive growth into the sacrum or the lumbosacral nerve roots indicating that surgery will never be possible even if substantial tumour down-sizing is seen.
* Presence of metastatic disease or recurrent rectal tumor.
* Familial Adenomatosis Polyposis coli (FAP), Hereditary Non-Polyposis Colorectal Cancer (HNPCC), active Crohn's disease or active ulcerative Colitis.
* Concomitant malignancies, except for adequately treated basal cell carcinoma of the skin or in situ carcinoma of the cervix uteri. Subjects with prior malignancies must be disease-free for at least 5 years.
* Known dihydropyrimidine dehydrogenase (DPD) deficiency.
* Any contraindications to MRI (e.g. patients with pacemakers)
* Medical or psychiatric conditions that compromise the patient's ability to give informed consent.
* Clinically significant (i.e. active) cardiac disease (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac dysrhythmia, e.g. atrial fibrillation, even if controlled with medication) or myocardial infarction within the past 12 months.
* Patients with known malabsorption syndromes or a lack of physical integrity of the upper gastrointestinal tract.
* Co-morbid illnesses or other concurrent disease which, in the judgment of the clinician obtaining informed consent, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens.
* Any investigational treatment for rectal cancer within the past year.
* Pregnancy or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Estimated)
Dates: Start 2017-11-23 (Actual); Primary Completion 2022-05-30 (Estimated); Study Completion 2025-11-23 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response rate (pCR). | 3 years
  pCR will be defined as the absence of viable tumor cells in the primary tumor and in the lymph nodes (ypT0N0) by histopathological assessment of the surgical specimen at the time of definitive rectal surgery.
3-year disease free survival (DFS) rate. | 3 years
  3-year DFS will be defined as the percentage of patients alive without recurrence of disease at 3 years measured from the date of randomization

SECONDARY OUTCOMES:
Overall survival (OS) | 5 years
  defined as the time from randomization to death from any cause
Radiological response by MRI imaging before surgery. | 3 years
Short and long-term toxicity. | 3 - 5 years
  According to common toxicology criteria of adverse events, version 3
Surgical complications. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Shereef E Mohammad, Principal Investigator — King Abdullah Medical City
Locations (1):
- King Abdullah Medical City, Holy Capital, Mecca, Makkah Western, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No